CLINICAL TRIAL: NCT06108206
Title: Adaptive Radiotherapy Based on Multi-Parametric Diffusion- and Perfusion-weighted Magnetic Resonance Imaging in Patients With Newly Diagnosed High-Grade Glioma
Brief Title: Adaptive Radiotherapy and MRIs Based on Patients With Newly Diagnosed High-Grade Glioma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Principal Investigator, Tony Jau Cheng Wang, Professor of Radiation Oncology (in Neurological Surgery), Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAU2309
Record Dates: First submitted 2023-10-23; First posted 2023-10-30 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma; Anaplastic Astrocytoma; Astrocytoma; Anaplastic Oligodendroglioma
Keywords: Adaptive Radiotherapy; High-grade glioma; Perfusion-weighted imaging; Diffusion weighted imaging
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Oligodendroglioma; Glioma

STUDY DESIGN:
Intervention Model Description: Adaptive Radiation to the Brain
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adaptive Radiotherapy (Experimental): Subjects will receive radiotherapy per standard of care over 30-33 once-daily fractions in addition to 7 brain MRIs each in every week of treatment. Subjects receiving hypofractionated radiotherapy will receive radiotherapy per standard of care over 15 once-daily fractions in addition to 4 brain MRIs each in every week of treatment.
  Interventions: Other: Adaptive Radiotherapy

INTERVENTIONS:
Other: Adaptive Radiotherapy — Each patient will undergo a brain MRI at the following time points:
  1. Baseline- within 2 weeks prior to the start of chemo-RT,
  2. Week #1- on Fractions # 4 or 5
  3. Week #2- between Fractions # 6-10 (at least 5 days after the Week 1 MRI)
  4. Week #3- between Fractions # 11-15 (at least 5 days after the Week 2 MRI)
  5. Week #4- between Fractions # 16-20 gadolinium contrast (at least 5 days after the Week 3 MRI)
  6. Week #5- on Fractions # 24 or 25 (after the start of the Conedown)
  7. Week #6- +/- 3 days of Fraction #30 (end of RT)
  Patients receiving hypofractionated radiotherapy will undergo a brain MRI at the following time points:
  1. Baseline- within 2 weeks prior to the start of your standard of care chemotherapy radiation treatment (chemo-RT),
  2. Week #1 - on Fractions #4 or 5
  3. Week #2 - between Fractions #6-10 (at least 5 days after the Week 1 MRI)
  4. Week #3 - between Fractions #11-15 (at least 5 days after the Week 2 MRI)

SUMMARY:
The purpose of this study is to find out if performing additional Magnetic Resonance Image (MRI) scans of the subjects' brain during each week of the radiation treatment of their high-grade glioma will help improve the radiation treatment.

DETAILED DESCRIPTION:
Diffusion weighted imaging (DWI) and Perfusion-weighted imaging (PWI) are validated MRI techniques that aid in diagnosis, prognosis, and assessment of treatment efficacy and, while they are utilized in select clinical settings, they have yet to make their way into routine clinical practice at most centers. DWI is a non-invasive MRI modality that has demonstrated an ability to predict for a response to radiation therapy in the primary treatment of patients with glioblastoma (GBM). PWI is one collection of measures that includes dynamic susceptibility contrast (DSC) enhancement and dynamic contrast-enhanced (DCE) imaging. The latter methods of MRI-adapted radiotherapy allow the opportunity to direct high-dose radiation to areas most likely to harbor resistant tumor while avoiding regions having a low likelihood of future recurrence. Multiple MRI sequences have been developed and validated that may identify high-risk areas in patients with High-grade glioma (HGG) and the ability to acquire multiple sequential time points creates an opportunity for dynamic radiotherapy that has not previously been explored. The current standard of care in radiotherapy does not incorporate any additional neuroimaging data.

This study hypothesizes that pre- and mid-treatment advanced imaging with (DWI) and (PWI) in patients with HGG can be used to generate an adaptive radiotherapy boost volume that correlates with areas of future recurrence and that this volume has a higher spatial correlation relative to the current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically proven diagnosis of glioblastoma, anaplastic astrocytoma, or anaplastic oligodendroglioma
* History and physical examination within 28 days prior to enrollment
* Karnofsky performance status 70 or greater
* Age 18 years or greater
* Negative pregnancy test for females of childbearing potential before 1st research MRI, performed in accordance to institutional guidelines.
* Plan to receive 59.4-60 Gy in 30-33 fractions of radiotherapy. Glioblastoma patients over 65 year-old can receive hypofractionated radiotherapy including 40 Gy in 15 fractions.

Exclusion Criteria:

* Prior therapy for tumor except for biopsy or resection, including prior radiotherapy to the brain.
* Clinical or radiological evidence of metastatic disease outside the brain
* Prior malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Prediction of progression of disease in patients with high-grade glioma. | 3 years
  To compare the volume of the current standard of care conedown volume definition with an MRI-based adaptive plan in predicting the location of disease progression in patients with high-grade glioma.

SECONDARY OUTCOMES:
Estimate the progression-free and overall survival in patient with high-grade glioma. | 3 years
  Assess the prognostic and predictive value of highly-diffusion weighted and perfusion-weighted imaging in estimating progression-free and overall survival in patients with high-grade glioma.

CONTACTS AND LOCATIONS:
Overall Officials: Tony J. Wang, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center/NYPH, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided